CLINICAL TRIAL: NCT04547218
Title: Study on Incidence of Elective Surgery Postponed During COVID-19 Pandemic in Geriatric Population
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Loh Pui San, Associate Professor, University of Malaya
Other Study IDs: 2020623-8801
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Age Problem; Surgery; Depression, Anxiety
Keywords: Geriatric population; COVID-19 pandemic; Elective surgery
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients: Above 65 year old patients undergoing elective surgery Inclusion criteria I. Geriatric patients ( age more than 65 y/o) II. All elective surgeries under GA
  Exclusion criteria I. Refuse to participate in the study II. Patients with cognitive disorders such as dementia and Alzheimer's disease

SUMMARY:
The COVID-19 pandemic has disrupted routine hospital services globally. The hospital services include surgeries for benign diseases, cancer surgery and obstetric surgery. A study conducted by CovidSurg Collaborative estimated that 28,404,603 operations would be cancelled or postponed during the peak 12 weeks of disruption due to COVID-19. Globally, 81.7% of benign surgery, 37.7% of cancer surgery and 25.4% of elective Caesarean sections would be cancelled or postponed. If countries increase their normal surgical volume by 20% post-pandemic, it would take a median 45 weeks to clear the backlog of operations resulting from COVID-19 disruption. This study aims to estimate total number of elective operations postponed during COVID-19 in geriatric population.

DETAILED DESCRIPTION:
An audit study will be conducted among geriatric patients that are admitted for elective surgeries in University Malaya Medical center (UMMC). Patients who fulfil inclusion/ exclusion criteria will be recruited with consent and will have a face-to-face interview in the surgical ward prior to their elective surgeries.

Data collection in the form of a questionnaire designed in English and filled up by the research interviewer is created to document patient demography, surgical details and level of depression/ anxiety prior to surgery.

The primary objective of this study is to find incidence of elective surgeries has postponed during COVID-19 pandemic in geriatric population. This overarching aim raises two secondary objectives of the research:

1. To find the incidents of cancer surgeries postponed during COVID-19 pandemic in geriatric population.
2. To find the physical and psychological impact of postponed elective surgery in geriatric population during COVID-19 pandemic.

Random convenience sampling will be conducted. Data will be collected using REDCap (Research Electronic Data Capture) system and analyzed using SPSS software. Results will be presented as mean ± standard deviation, median or frequency (percentages) as appropriate. Mann-Whitney U test will be used for non-normally distributed data while t test will be used for normally distributed data. The qualitative data analysis will be performed using chi-square test or Fisher's exact test if insufficient numbers are present. A p value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients (aged 65 and above)
* All elective surgeries under general anesthesia, regional anesthesia and ALA

Exclusion Criteria:

* Refuse to participate in the study
* Patients with cognitive disorders such as dementia and Alzheimer's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric population undergoing elective surgery during COVID-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of elective surgeries has postponed during COVID-19 pandemic in geriatric population | June 2020 - October 2020
  The frequencies of diagnosed surgical indication before pandemic but surgeries deferred until re-opening of full elective lists will be documented.

SECONDARY OUTCOMES:
Incidence of cancer surgeries postponed during COVID-19 pandemic in geriatric population | June 2020 - December 2020
  The frequencies of diagnosed malignant cases with surgical indication before pandemic but surgeries deferred until re-opening of full elective lists will be documented.
Physical and psychological impact of postponed elective surgery in geriatric population during COVID-19 pandemic | June 2020 - December 2020
  Two scores will be used:
  1. The Hospital Anxiety and Depression Scale (HADS) with response in a 4-point scale (from 0 to 3) referring to overt symptoms within the last week. The total score for each component ( anxiety and depression) will be summed up to give an outcome such as 0-7 normal, 8-10 borderline abnormal and 11- 21 as abnormal.
  2. SF-36 with 36 questions to cover eight domains of health.
     1. Limitations in physical activities.
     2. Limitations in social activities
     3. Limitations in usual role activities
     4. Bodily pain
     5. General mental health (psychological distress and well-being)
     6. Limitations in usual role activities
     7. Vitality (energy and fatigue)
     8. General health perceptions Eight scaled scores with each directly transformed into a 0-100 scale, lower scores mean more disabiity.

CONTACTS AND LOCATIONS:
Overall Officials: Pui San Loh, FANZCA, Principal Investigator — Department of Anesthesiology & Intensive Care, University of Malaya
Locations (1):
- Department of Anesthesiology & Intensive Care, Faculty of Medicine, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] COVIDSurg Collaborative. Elective surgery cancellations due to the COVID-19 pandemic: global predictive modelling to inform surgical recovery plans. Br J Surg. 2020 Oct;107(11):1440-1449. doi: 10.1002/bjs.11746. Epub 2020 Jun 13. PMID 32395848
- [Background] University of Birmingham and College of Surgeons, Academy of Medicine of Malaysia news release. COVID-19 patients who undergo surgery are at increased risk of postoperative death - global study.
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230